CLINICAL TRIAL: NCT05309629
Title: An Open-label Phase 2 Study of QL1706 Plus Carboplatin and Etoposide as First-line Treatment in Patients With Extensive-stage Small Cell Lung Cancer
Brief Title: Safety and Efficacy Study of First-line Treatment With QL1706 Plus Chemotherapy in Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-209
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2022-11

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706+chemotherapy (Experimental): Participants received intravenous infusions of QL1706 5mg/kg in combination with carboplatin to achieve an initial target area under the concentration-time curve (AUC) of 5 mg/mL/min followed by etoposide 100 mg/m^2 on Day 1 of every 21-day cycle for 4-6 cycles. On Days 2 and 3 of every 21-day cycle, etoposide 100 mg/m^2 was administered alone for 4-6 cycles. Thereafter, participants received maintenance QL1706 5mg/kg on Day 1 of every 21-day cycle until progressive disease, intolerable toxicity, withdrawal of consent, death, or study termination by the Sponsor.
  Interventions: Drug: QL1706; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: QL1706 — Intravenous infusions of QL1706 5mg/kg on Day 1 of every 21-day cycle.
Drug: Carboplatin — Carboplatin intravenous infusion to achieve an initial target AUC of 5 mg/mL/min was administered on Day 1 of each 21-day cycle for 4-6 cycles.
Drug: Etoposide — Etoposide intravenous infusion was administered at a dose of 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for 4-6 cycles.

SUMMARY:
This is an open label, phase 2 clinical study to evaluate the safety, tolerability, efficacy, pharmacokinetic (PK) profile, and immunogenicity of QL1706 plus carboplatin and etoposide as first-line therapy in patients with extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate voluntarily and sign informed consent.
2. Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system)
3. No prior systemic treatment for ES-SCLC
4. Eastern Cooperative Oncology Group performance status of 0 or 1
5. Measurable disease, as defined by RECIST v1.1
6. Adequate hematologic and end organ function

Exclusion Criteria:

1. Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation
2. Active, known or suspected autoimmune disease
3. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, radiation pneumonia requiring steroid treatment or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
4. Positive test result for human immunodeficiency virus (HIV)
5. Active hepatitis B or hepatitis C
6. Significant cardiovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced At Least One Adverse Event (AE) | Up to approximately 2 years
  An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants who experienced at least one AE is presented.

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response (OR) | Up to approximately 2 years
  The efficacy outcome of objective response rate (ORR) as assessed by the investigator using RECIST v1.1
Duration of Response (DOR) | Up to approximately 2 years
  The efficacy outcome of DOR as assessed by the investigator using RECIST v1.1
Duration of Progression-Free Survival (PFS) | Up to approximately 2 years
  The efficacy outcome of PFS as assessed by the investigator using RECIST v1.1
Duration of Overall Survival (OS) | Up to approximately 2 years and a half
  Baseline until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China